CLINICAL TRIAL: NCT04735939
Title: Chronotherapy for Radiotherapy of Glioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: xhechun5
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: To Determine Whether the Timing of Radiotherapy Has an Effect on Patient Outcomes
Keywords: radiotherapy, glioma, outcomes
MeSH Terms: conditions — Glioma | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- morning dosing radiotherapy
  Interventions: Radiation: radiotherapy
- evening dosing radiotherapy
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — Determine whether there is a difference in outcomes seen when patients are assigned to take their radiotherapy at either a morning time or evening time.

SUMMARY:
This study aims to determine if there is any difference in the efficacy of radiotherapy for glioma outcomes in the morning or in the evening. The study team believes that there may be a benefit to taking the radiotherapy at a certain time of day. To test this theory the study asks participants who are already taking radiotherapy for glioma consistently at either the morning or in the evening based on when they currently take their radiotherapy. There will be this study visits where the participant will be asked to fill in questionnaires related to their neurological symptoms, their sleep habits, sleep quality, survival situation, and general health information followed by a blood draw.

DETAILED DESCRIPTION:
The objective of this study is to determine whether the timing of radiotherapy to treat glioma has an effect on patient outcomes.

Primary objective: Determine whether there is a difference in outcomes seen when patients are assigned to take their radiotherapy at either a morning time or evening time.

The Investigator hypothesize that administration time of radiotherapy during the day can affect the clinical outcomes in glioma patients.

Specific Aims Include:

* Determine whether morning vs. evening dosing radiotherapy could affect the survival time of glioma patients.
* Determine whether morning vs. evening dosing radiotherapy could affect the KPS score of glioma patients.
* Determine whether morning vs. evening dosing radiotherapy could affect the cognitive function of glioma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Pathological or cytological diagnosis of glioma;
3. Normal liver and kidney function.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Second primary malignancy;
3. Severe lung infection;
4. with high blood pressure although treated with medication;
5. Patients with myocardial ischemia or myocardial infarction, arrhythmia (including QT interval > 440 ms) or grade II cardiac insufficiency;
6. Arteriovenous thrombosis in 6 months prior to first administration, Such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism;
7. Serious heart, lung and bone marrow impairment;
8. History of severe hypertension or cerebral hemorrhage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be divided into two groups.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
survival time of glioma patients | 1/1/2021-31/12/2021
  Determine whether morning vs. evening dosing radiotherapy could affect the survival time of glioma patients.

SECONDARY OUTCOMES:
KPS score of glioma patients. | 1/1/2021-31/12/2021
  Determine whether morning vs. evening dosing radiotherapy could affect the KPS score of glioma patients.

OTHER OUTCOMES:
cognitive function of glioma patients | 1/1/2021-31/12/2021
  Determine whether morning vs. evening dosing radiotherapy could affect the cognitive function of glioma patients.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No